CLINICAL TRIAL: NCT03507621
Title: Comparison of the Postoperative Pain Scores and of the Neuroendocrine Stress Responses of Blood and Follicular Fluid of Two Different Anesthesia Methods in Oocyte Pick up Applications
Brief Title: Sevoflurane Versus Propofol; Neuro Endocrine Response in Patients of Oociyt Pick up
Status: Completed | Type: Observational
Sponsor: Yavuz Orak (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Sponsor-Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Other Study IDs: 2017/12-16
Record Dates: First submitted 2018-02-22; First posted 2018-04-25 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia; Infertility; Pain, Postoperative; Stress, Psychological
MeSH Terms: conditions — Infertility; Pain, Postoperative; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol Group: 1- Propofol Group: Propofol group will use 1 mg / kg propofol for the patient.Preoperative blood will be taken from the patients and cortisol, acth, glucagon, aldosterone, adrenalin, noradrenalin, PGE2, CRH will be studied. During the operation, the patient's systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, oxygen saturation will be followed. Analgesia will be provided according to the body movements of the patient and VAS measurement will be performed. Remifentanyl will be used as a anelgesic 0.5 mcg/ kg during operation. The patient's pain will be assessed by the VAS (Visuel Analogue Scale) scoring system and during the first hour postoperatively after the patient's consciousness is complete .
- Sevoflurane Group: 1- Sevofluran Group: sevoflurane was administered at one minimum alveolar concentration (MAC) to end-tidal concentrations of 3% to 5%.Preoperative blood will be taken from the patients and cortisol, acth, glucagon, aldosterone, adrenalin, noradrenalin, PGE2, CRH will be studied. During the operation, the patient's systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, oxygen saturation will be followed. Analgesia will be provided according to the body movements of the patient and VAS measurement will be performed. Remifentanyl will be used as a anelgesic 0.5 mcg/ kg during operation. The patient's pain will be assessed by the VAS (Visuel Analogue Scale) scoring system and during the first hour postoperatively after the patient's consciousness is complete.

SUMMARY:
Patients in the study will be grouped as 1st group Propofol, 2nd Group Sevofluran.Preoperative blood will be taken from the patients and cortisol, acth, glucagon, aldosterone, PGE2, CRH will be studied. During the operation, the patient's systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, oxygen saturation will be followed. Analgesia will be provided according to the body movements of the patient and VAS measurement will be performed. The patient's pain will be assessed by the VAS (Visuel Analogue Scale) scoring system and during the first hour postoperatively after the patient's consciousness is complete . Hormones such as cortisol, acth, glucagon, aldosterone, PGE2, CRH will be studied biochemically in the follicular fluid and blood of the patient postoperatively. The aim of in the study is to compare the effect of propofol and sevoflurane routinely applied in IVF centers on postoperative pain scores and stress hormones in blood and follicular fluid in a painful and stressful application of egg collection

DETAILED DESCRIPTION:
In vitro fertilization (IVF) is the technique that allows male and female sperm and egg fertilization to occur outside the female body, and is the most common assisted reproductive technique. Collection of eggs (oocytes) from female ovaries is called oocyte pick-up (OPU) in the process. Initially started to be implemented towards the end of 1970. In the last 30 years, the number of infertile couples has been increasing and trying to have children with in vitro fertilization techniques. Different anesthetic agents are used for the oocyt pick-up procedure. Studies have shown that anesthetic agents are detected in follicular fluid. Animal and human studies indicate that anesthetic agents may negatively affect the development of oocytes and embryos. However, the possible effects of anesthetic drugs on oocyte physiology and embryo development have not yet been sufficiently investigated. Currently, the possible effects of different anesthetic agents on the oocyte are discussed. In one study, the highest number of oocytes per patient and the lowest number of mature oocytes in the thiopental sodium and sevoflurane groups were determined. On the other hand, there are studies showing a marked increase in 1PN and 3PN oocytes when there is a decrease in normal fertilized oocytes in the propofol group. These results suggest that oocyte cytoskeleton may be an effect of propofol. It is known that propofol is detected in human follicular fluid. In addition, harmful effects on division and fertilization were shown in mouse models. Despite this, propofol is one of the most commonly used agents. In another study showed that , sevoflurane has a genotoxic effect on hamster ovay cell. However, when another group performed the same tests to test propofol genotoxicity effects were not found. Patients feel anxiety before oocyte processing, and sometimes feel severe pain during the procedure. Surgical procedures and interventional procedures applied to the disease are characterized by pain, neurohumoral, immunologic, metabolic changes resulting in a complex stress response. The magnitude of the resulting stress response depends on various factors such as the severity and duration of the surgical trauma, patient age, peroperative and postoperative pain, anesthetic method and surgical technique. Even if adequate analgesia is provided in the egg collection process, the patients usually feel pain in the peroperative and postoperative period. It has been reported that these changes induced by stress in the literature may lead to complications in perioperative and postoperative period. Many studies in the literature have indicated that the choice of anesthetic agent may affect stress response by stimulating, inhibiting, and alleviating pathophysiological pathways leading to neurohumoral and immunological changes. The effects of sevoflurane and propofol anesthesia on the surgical trauma on the neurohumoral response have been investigated, but some aspects have not yet been clarified. Patients in the study will be grouped as 1st group Propofol, 2nd Group Sevofluran.Preoperative blood will be taken from the patients and cortisol, acth, glucagon, aldosterone, PGE2, CRH will be studied.During the operation, hemodynamics (systolic blood pressure, diastolic blood pressure, heart rate, mean arterial pressure, oxygen saturation) will be recorded during the operation at 1,3,5,7,10,15 minutes. Additional analgesic and anesthesia requirements and body movements will be recorded during the operation. Analgesia will be provided according to the body movements of the patient and VAS measurement will be performed. The patient's pain will be assessed by the VAS (Visuel Analogue Scale) scoring system and hemodynamic parameters (systolic blood pressure, diastolic blood pressure, heart rate, mean arterial pressure, oxygen saturation) during the first hour (1 mınute,5. minute, 15. minute,30. minute, 60. minute) postoperatively after the patient's consciousness is complete .Analgesic (Naproxen Sodium) will be administered when the pain score (VAS) is 5 or greater than 5. Hormones such as cortisol, acth, glucagon, aldosterone, PGE2, CRH will be studied biochemically in the follicular fluid and blood of the patient postoperatively. The aim of the study is to compare the effect of propofol and sevoflurane routinely applied in IVF centers on postoperative pain scores and stress hormones in blood and follicular fluid in a painful and stressful application of egg collection. In this study, two different anesthetic agents administered with propofol and sevoflurane will be used to compare the peroperative analgesic consumption and postoperative pain levels. At the same time, it will be determined which anesthetic agent is suitable for oocyte collection by looking at the neurohumoral stress hormones in blood and follicular fluid. The findings will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old and under 40 years old
* Volunteers who want to participate in the work

Exclusion Criteria:

* Patients under 18 and over 40
* Those who do not want to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients between the ages of 18 and 40 who have undergone IVF practice constitute the patient population.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
preoperative and postoperative neuroendocrine stress hormones in blood | baseline about ten minutes before operatİon ,and Change from baseline about ten minutes after operation
  To evaluate the impact on the circulating levels of kortizol mikrogram/dl, acth pg/ml, glukagon pg/ml,aldosteron pg/ml, PGE2 pg/ml, CRH ng/ml
Pain Scores | after the operation in 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes.Each unit will be evaluated separately within itself
  VAS (Visuel Analogue Scale) . Score from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated
postoperative neuroendocrine stress hormones in follicular fluid | Change from baseline about ten minutes after operation
  kortizol mikrogram/dl, acth pg/ml, glukagon pg/ml, aldosteron pg/ml, PGE2 pg/ml, CRH ng/ml

SECONDARY OUTCOMES:
Hemodynamics and oxygen follow-up | During the operation, 1 minute, 3 minutes, 5 minutes, 7 minutes, 10 minutes, 15 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, oxygen saturation
Hemodynamics and oxygen follow-up | after the operation in 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate,

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz orak, md, Study Director — Kahramanmaraş Sutcu Imam University Faculty of Medicine Kahramanmaraş/ Turkey
Locations (1):
- Kahramanmaras Sutcu Imam Univercity Faculty of edicine, Kahramanmaraş, Onikişubat, Turkey (Türkiye)